CLINICAL TRIAL: NCT03320096
Title: Evaluation of the Ulthera System for Treating Axillary Hyperhidrosis
Acronym: ULT-218
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M960001007; DRKS00011603 (Registry Identifier: DRKS)
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Results first posted 2019-07-10 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2017-10

CONDITIONS: Axillary Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microfocused ultrasound with visualization (Experimental)
  Interventions: Device: Microfocused ultrasound with visualization

INTERVENTIONS:
Device: Microfocused ultrasound with visualization — Subjects will receive 2 treatments (day 1 and day 30), each at a 3.0mm depth and 0.30 Joule of energy. Treatment will be delivered in a 3*4 grid, 12 treatment squares, delivering 60 lines of treatment per square, i.e., 720 lines per axilla in each treatment (1440 lines total per treatment.)
  Other Names: Ultherapy; Ulthera treatment

SUMMARY:
To evaluate the Ulthera System and the 7-3.0mm transducer for treating axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75 years.
* Diagnosis of bilateral axillary hyperhidrosis refractory to previous topical therapies.
* At least 50 mg of spontaneous resting axillary sweat production in each axilla measured gravimetrically at room temperature/humidity (20 - 25.6°C/20-80%) over a period of 5 minutes. (Patients should be at rest for at least 30 minutes after physical exercise including walking.)
* HDSS score of 3 or 4. An attempt will be made to approximate an equal number of scores 3 and 4.
* Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID, and Vitamin E in the 2 weeks prior to each study treatment .

Exclusion Criteria:

* Dermal disorder including infection at anticipated treatment sites in either axilla.
* Previous botulinum toxin treatment of the axilla in the past year.
* Expected use of botulinum toxin for the treatment of any other disease during the study period.
* Known allergy to starch powder, iodine, lidocaine, or epinephrine.
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (2):
- Germany (2):
  - Rosenpark Research, Study Research Center; Merz Investigational Site #0490099, Darmstadt
  - Haut- & Laserzentrum, Merz Investigational Site #0490362, Potsdam

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites in Germany.
Pre-assignment Details: A total of 20 participants were screened, enrolled and treated in the study.
Groups:
- Ultherapy Treatment: Participants received two dual-depth Ultherapy treatment to each axilla at a treatment depth of 3.0 millimeter (mm) using 7-megahertz (MHz) transducer with 0.30 joules (J) of energy on Days 0 (Treatment 1) and 30 (Treatment 2). Participants were administered treatment in 3 inch*4 inch grid, in at least 12 treatment squares. At each treatment visit, participants received a minimum of 720 treatment lines to each axilla (minimum of 1440 total lines of treatment for both axillae), delivering 60 treatment lines per treatment square.
Period: Overall Study
Arm/Group | Ultherapy Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was the subset of participants in the safety evaluation set (SES) for whom the primary efficacy variable was available (that is, all participants who had baseline and at least one post-baseline value of the primary efficacy variable). SES was the subset of all participants who were exposed to study treatment at least once.
Groups:
- Ultherapy Treatment: Participants received two dual-depth Ultherapy treatment to each axilla at a treatment depth of 3.0 mm using 7-MHz transducer with 0.30 J of energy on Days 0 (Treatment 1) and 30 (Treatment 2). Participants were administered treatment in 3 inch*4 inch grid, in at least 12 treatment squares. At each treatment visit, participants received a minimum of 720 treatment lines to each axilla (minimum of 1440 total lines of treatment for both axillae), delivering 60 treatment lines per treatment square.
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 20
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.1 (4.0)
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Skin Type I | 0
    Skin Type II | 15
    Skin Type III | 4
    Skin Type IV | 1
    Skin Type V | 0
    Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hyperhidrosis Disease Severity Scale (HDSS) Score Reduction at Day 30 Post Second Treatment
Description: Treatment success was defined as a reduction on the HDSS score from a value of 3 or 4 at baseline to a 1 or 2 at 30-day post second treatment. The HDSS was a validated scale used for primary axillary/underarm hyperhidrosis participants. HDSS provides a qualitative measure of the severity of participant's condition based on how it affects their daily activities. It is a 4-point scale (1-4) with scores as: 1 (underarm sweating was never noticeable and never interferes with daily activities); 2 (underarm sweating was tolerable but sometimes interferes with daily activities); 3 (underarm sweating was barely tolerable and frequently interferes with daily activities); and 4 (underarm sweating was intolerable and always interferes with daily activities).
Time Frame: Day 60 (30 days post second treatment)
Population: All evaluable treated participants in FAS who received a complete or partial study treatment and completed a follow-up visit at Day 30 post second treatment. The FAS was the subset of participants in SES for whom primary efficacy variable was available. The SES was the subset of all participants who were exposed to study treatment at least once.
Measure: Number; unit: participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 20
participants | 11

2. Secondary Outcome: Number of Participants With HDSS Score Reduction at Day 90 Post Second Treatment
Description: Treatment success was defined as an HDSS score reduction from a value of a 3 or 4 to a 1 or 2 at 90-day post second treatment. The HDSS was a validated scale used for primary axillary/underarm hyperhidrosis participants. HDSS provides a qualitative measure of the severity of participant's condition based on how it affects their daily activities. It is a 4-point scale (1-4) with scores as: 1 (underarm sweating was never noticeable and never interferes with daily activities); 2 (underarm sweating was tolerable but sometimes interferes with daily activities); 3 (underarm sweating was barely tolerable and frequently interferes with daily activities); and 4 (underarm sweating was intolerable and always interferes with daily activities).
Time Frame: Day 120 (90 days post second treatment)
Population: The FAS was the subset of participants in the SES for whom the primary efficacy variable was available (that is, all participants who had baseline and at least one post-baseline value of the primary efficacy variable). The SES was the subset of all participants who were exposed to study treatment at least once.
Measure: Number; unit: participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 20
participants | 15

3. Secondary Outcome: Number of Participants With Gravimetric Axillary Sweat Reduction by at Least 50 Percent (%) at Days 30 and 90 Post Second Treatment
Description: Treatment success for gravimetric sweat production test was defined as a 50% or more reduction in spontaneous sweat production compared to baseline at 30 days and 90 days post second treatment. Gravimetric sweat production was measured using a pre-weighed filter paper placed into the axilla for a period of 5 minutes. The paper was removed and weighed and rate of sweat production was calculated in milligram per 5 minute (mg/5 min) based on the difference in end-weight and pre-weight.
Time Frame: Days 60 (30 days post second treatment) and 120 (90 days post second treatment)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 20
participants
  Day 60 | 12
  Day 120 | 15

4. Secondary Outcome: Number of Participants Who Showed Improvement With the Starch Iodine Test at Days 30 and 90 Post Second Treatment
Description: Improvement for the starch iodine test was defined as a reduction in the dark blue starch iodine area, both the left and right axilla needed to show improvement for a participant to be classified as improved. The starch iodine test was used to assess the area involved in excessive sweating by visually identifying areas that were actively producing sweat. The test was performed by applying iodine solution to the axilla and allowing the solution to dry. After drying, starch was sprinkled on the area. The light-brown iodine color turns dark purple as iodine-starch complexes form in the liquid medium with the sweat rising to the surface of the affected area. Starch iodine test was captured with digital images.
Time Frame: Days 60 (30 days post second treatment) and 120 (90 days post second treatment)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 20
participants
  Day 60 | 16
  Day 120 | 20

ADVERSE EVENTS:
Time Frame: Baseline up to Day 120
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Ultherapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 18/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultherapy Treatment (N=20)
Headache (Nervous system disorders) | 2
Tingling (Nervous system disorders) | 8
Hematoma (General disorders) | 16
Tenderness (General disorders) | 3
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neuritis (Nervous system disorders) | 1
Swelling (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/96/NCT03320096/Prot_SAP_000.pdf